CLINICAL TRIAL: NCT03590028
Title: An Early Real-Time Electronic Health Record Risk Algorithm for the Prevention and Treatment of Acute Kidney Injury: A Randomized Trial of an Early Standardized, Personalized Nephrology Intervention
Brief Title: An Early Real-Time Electronic Health Record Risk Algorithm for the Prevention and Treatment of Acute Kidney Injury
Acronym: ESTOP-AKI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-1081
Record Dates: First submitted 2018-06-21; First posted 2018-07-18 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Nephrology Consult (ENC) (Experimental): The ENC will be a structured consultative note that will provide detailed recommendations around issues such as Differential Diagnosis, Drug Dosing and Volume Status. The research ENC will have a daily follow-up with documented recommendations.
  Interventions: Other: Early Nephrology Consult (ENC)
- Standard of Care (SOC) (Active Comparator): Subjects will receive nephrology consultation at the typical timepoint after symptoms of AKI appear.
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Other: Early Nephrology Consult (ENC) — The electronic risk prediction algorithm (ESTOP-AKI) will interface with electronic medical data to determine the likelihood for the patient to develop AKI. Early Nephrology Consult (ENC) will be implemented. A nephrologist will assess the subject and consult with their care team to advise a treatment plan during the hospitalization.
  Arms: Early Nephrology Consult (ENC)
Other: Standard of Care (SOC) — Subjects will receive nephrology consultation at the typical timepoint after symptoms of AKI appear.
  Arms: Standard of Care (SOC)

SUMMARY:
This is a single center randomized trial that seeks to determine if the use of an automated real-time electronic medical record Acute Kidney Injury (AKI) risk score can improve patient outcomes through the use of an early standardized nephrology focused intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old
2. Initial ESTOP AKI score ≥0.01 within the last 8 hours.

Exclusion Criteria:

1. Voluntary refusal or missing written consent of the patient / legal representative.
2. Patients with a known history of end-stage renal disease on dialysis (including renal transplantation).
3. Patients without a measured serum creatinine value during their inpatient stay.
4. Patients with a creatinine >4.0 mg/dl at the time of admission or available in the electronic health record (EHR) from the last 6 months.
5. Patients with prior episode of Kidney Disease Improving Global Outcomes (KDIGO) defined AKI during this same hospitalization- regardless of ESTOP AKI score.
6. Patients with prior renal consultation during their admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Peak change in milligrams per deciliter (mg/dL) in serum creatinine (SCr) level over a 7-day interval | 7-day interval
  The primary endpoint of interest, change in serum creatinine (SCr), is the peak change from study entry in SCr level over a 7-day interval. The change in SCr is defined as the maximal change in creatinine over this interval, and aim to detect a clinical difference in change in SCr between the SOC and ENC treatment groups.

OTHER OUTCOMES:
Differences by treatment group in the proportion by percent and time in days to specified medical events. | 3 months
  The differences will be measured by treatment group in the proportion and time to event of patients who a) develop > Stage 2 AKI, b) require renal replacement therapy (RRT), c) undergo intensive care unit (ICU) transfer, and/or d) require non-research nephrology consult.
Comparison of treatment groups in the proportion by percent and time in days of length of stay (LOS) in the hospital. | 3 months
  The differences will be measured by treatment group in the proportion by percent and time in days of LOS in the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Koyner, MD, Principal Investigator — University of Chicago Medicine
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koyner JL, Martin J, Carey KA, Caskey J, Edelson DP, Mayampurath A, Dligach D, Afshar M, Churpek MM. Multicenter Development and Validation of a Multimodal Deep Learning Model to Predict Moderate to Severe AKI. Clin J Am Soc Nephrol. 2025 Apr 15;20(6):766-778. doi: 10.2215/CJN.0000000695. PMID 40232856